CLINICAL TRIAL: NCT02724059
Title: The Role of Endobronchial Ultrasound Elastography in the Diagnosis of Mediastinal Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Adel Salah Bediwy, Professor, Tanta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TFMEC221015
Record Dates: First submitted 2016-03-19; First posted 2016-03-31 (Estimated); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Mediastinum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients with mediastinal lesions (Experimental): Endo bronchial ultrasound (EBUS) with elastography followed by TBNA
  Interventions: Procedure: EBUS with elastography followed by TBNA

INTERVENTIONS:
Procedure: EBUS with elastography followed by TBNA — Endo bronchial ultrasound (EBUS) with elastography followed by TBNA from mediastinal lesions or lymph nodes

SUMMARY:
The study will include 30 patients with hilar/mediastinal lymph nodes detected by thoracic CT either there was a known lung malignancy (for staging purpose) or not (for diagnosing purpose).

All patients will undergo to EBUS-guided TBNA. Elastography will be performed on all lymph nodes that will be candidates for EBUS TBNA. Mediastinoscopy or other invasive procedures will be performed if EBUS-guided TBNA doesn't provide representative material.

DETAILED DESCRIPTION:
All patients will be subjected to the following parameters:

1. Thorough history taking and full clinical examination.
2. Chest X-ray (postro-anterior and lateral views) before and after the procedure.
3. Recent Computed Tomography (CT chest) with contrast.
4. Laboratory studies:

   * Complete liver functions.
   * Blood urea and serum creatinine.
   * Complete blood picture (including platelet count).
   * Erythrocyte sedimentation rate (ESR).
   * Fasting and postprandial blood sugar.
5. Preoperative evaluation: Pulmonary function tests (PFT), Electrocardiogram (ECG), arterial blood gases (ABG) and coagulation profile (including bleeding & clotting times, prothrombin time& activity and activated partial thromboplastin time (APTT)) and oral anticoagulants should be stopped before the procedure for at least 48 hours.
6. Color doppler ultrasound in suspected vascular lesions.
7. Clinical and radiological follow up of patients over 1 week after the procedure to detect the occurrence of any complications.
8. The biopsy samples will be examined histopathologically. EBUS-guided TBNA examinations will be performed in all cases at the pulmonary department of Tanta University Educational Hospital as an outpatient procedure in a dedicated bronchoscopy suit with Pantex EBUS probe and Hitachi ultrasound a 7.5 MHz, BF-UC160F (Olympus Optical Co., Tokyo, Japan, approved by FDA) convex probe bronchoscope and EU C2000 processor (Olympus, Tokyo, Japan) by oral route and in the supine position under local anesthesia with lidocaine and conscious sedation with intravenous midazolam.

Lymph nodes will be identified according to the Mountain's regional lymph node classification system (5). The lymph node stations of 2, 4, 7, 10 and 11 will be evaluated systematically. After the appearance of target lymph nodes, the diameter, shape, edge definition, internal echo distribution, and location of the lymph nodes will be recorded in conventional B mode by ultrasound.

Elastography will be performed on all lymph nodes that will be candidates for EBUS TBNA. The scan range will include the entire lymph node and the surrounding normal tissue. Elastographic and B mode images will be simultaneously displayed side by side on the monitor. Elastographic patterns will be described according to the dominant colors and their distribution within the target lymph node. The strain ratio can be only measured when good contact and appropriate compression of the transducer will be achieved, as indicated by the elastography image on the ultrasound processor. The largest possible area of the node will be outlined from the superimposed elastography image; the same procedure will be performed on a similar-sized area that is surrounded by apparently normal tissue. The ultrasound processor measured the strain of each area as a quantitative figure, and the strain ratio between the two areas will be calculated. The strain ratio will be recorded a minimum of 3 times prior to EBUS-TBNA. The means of these recordings will also be calculated. (4) After elastography, EBUS TBNA will be performed with a Cook 22 gauge needle (c976006, Cook Ireland Limited Liability Company, Ireland). The number of passes per patient will be recorded. N3 nodes will be sampled first and then N2 nodes to avoid contamination in lung cancer patients. Histological and cytological specimens will be collected and sent to the laboratory for subsequent analysis by pathologist who will be blinded to the elastography values.

Aspiration specimen will be considered "insufficient" if there will not be an adequate number of lymphocytes on the smear. A definitive diagnosis of malignancy from the EBUS TBNA specimens will be considered a positive result. No clear evidence of malignancy or inadequate specimen by EBUS TBNA will be deemed a negative result.

For the patients whose results are negative for malignancy, more invasive procedures such as mediastinoscopy will be done to confirm the diagnosis or radiologic follow-up on the outcome of the LNs for at least 6 months. On follow-up, LNs that persisted in size, diminished, or resolved will be considered benign. A diagnosis of tuberculosis or sarcoidosis will be made based on cytopathology that showed the presence of caseating or noncaseating granuloma, in addition to clinical, radiological, and microbiological findings.

ELIGIBILITY:
Inclusion Criteria:

* Hilar/mediastinal lymph nodes with a short axis more than 1 cm on thoracic CT scan and/or PET-CT suspicious for malignancy with or without known lung malignancy.
* Hilar and/or mediastinal lymph nodes positive on PET/CT scan without regarding the diameter suspicious for malignancy.
* Recurrence or restaging of NSCLC after chemotherapy or radiation.
* Diagnosis of both benign and malignant mediastinal lesions.

Exclusion Criteria:

* Cardiovascular instability.
* Lack of patient cooperation, e.g. intractable cough, inability to remain motionless or altered consciousness.
* Bleeding diathesis (activated partial thromboplastin time (APTT) ratio or international normalized ratio (INR) <1.3 or platelet count of <50000 per mm3).
* Border line respiratory failure and patient on mechanical ventilation.
* Severe chronic obstructive pulmonary disease (COPD) (FEV1<1 liter or <35% predicted).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2015-11; Primary Completion 2016-04 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with correct diagnosis of mediastinal lesions (benign or malignant) using elastography | 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Adel S Bediwy, MD, Study Chair — Chest Department, Faculty of Medicine, Tanta University; Mohamed S Hantera, MD, Principal Investigator — Chest Department, Faculty of Medicine, Tanta University; Ayman El-Saqa, MD, Principal Investigator — Pathology Department, Faculty of Medicine, Tanta University; Dalia ElSharawy, MD, Principal Investigator — Chest Department, Faculty of Medicine, Tanta University
Locations (1):
- Chest Department, Faculty of Medicine, Tanta University, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Jiang JH, Turner JF Jr, Huang JA. Endobronchial ultrasound elastography: a new method in endobronchial ultrasound-guided transbronchial needle aspiration. J Thorac Dis. 2015 Dec;7(Suppl 4):S272-8. doi: 10.3978/j.issn.2072-1439.2015.12.53. PMID 26807274